CLINICAL TRIAL: NCT07262619
Title: A Multicenter, Multi-Part, Phase 1/2 Study of EIK1005 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors, Including Checkpoint Inhibitor Naïve Participants With Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) Tumors
Brief Title: EIK1005-002: A Clinical Research Study Evaluating EIK1005, a Werner Helicase Inhibitor, as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors Including Microsatellite Instability High (MSI-H) Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EIK1005-002
Record Dates: First submitted 2025-11-10; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors; MSI-H or dMMR Advanced Solid Tumors; MSI-H/dMMR Gastric Cancer; MSI-H/dMMR Colorectal Cancer; MSI-H/dMMR Gastroesophageal-junction Cancer; Endometrial Cancer; Mismatch Repair Deficient or MSI-High Solid Tumors
Keywords: Werner helicase; WRN; MSI-H; dMMR; DNA mismatch repair; EIK1005; Advanced Solid Tumors; Metastatic; MSI-H/dMMR Endometrial Cancer; MSI-H/dMMR Prostate Cancer; Pembrolizumab; Mismatch Repair Deficient (dMMR); Microsatellite Instability High (MSI-H)
MeSH Terms: conditions — Endometrial Neoplasms; Turcot syndrome; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A (Dose escalation, Monotherapy) (Experimental): EIK1005 will be given as monotherapy in participants without alternative treatment options.
  Interventions: Drug: EIK1005
- Part 1B (Dose escalation, Combination with pembrolizumab) (Experimental): EIK1005 will be given in combination with pembrolizumab to participants with Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) solid tumors.
  Interventions: Drug: EIK1005; Drug: Pembrolizumab (KEYTRUDA® )
- Part 2 (Dose optimization, Monotherapy) (Experimental): Participants with Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) advanced solid tumors will be randomized to receive EIK1005 monotherapy at one of the two identified doses selected from Part 1A.
  Interventions: Drug: EIK1005

INTERVENTIONS:
Drug: EIK1005 — EIK1005 is a selective inhibitor of the Werner helicase.
Drug: Pembrolizumab (KEYTRUDA® ) — Pembrolizumab is a PD-1 inhibitor.
  Arms: Part 1B (Dose escalation, Combination with pembrolizumab)

SUMMARY:
The goal of this clinical trial is to determine the most effective dose of EIK1005 that a person can take safely. Additionally, this study will test how well EIK1005 is tolerated alone and in combination with pembrolizumab in treating patients with advanced cancer.

DETAILED DESCRIPTION:
This Phase 1/2 study (EIK1005-002) will investigate the safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of EIK1005 as a monotherapy and in combination with pembrolizumab in participants with advanced solid tumors, including participants with Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) Tumors.

The study will be conducted in 2 parts: Part 1 and Part 2, with Part 1 being further divided into Part 1A and Part 1B as described below:

* Part 1A (monotherapy dose escalation): participants will receive EIK1005 only.
* Part 1B (combination dose escalation): participants will receive EIK1005 in combination with pembrolizumab.
* Part 2 (dose optimization): participants will be randomized 1:1 to monotherapy with EIK1005 at one of the two selected doses from Part 1A to identify the dose of EIK1005 in monotherapy for subsequent studies.

ELIGIBILITY:
Key Inclusion Criteria:

1. is ≥ 18 years of age at the time of signing the informed consent.
2. has a life expectancy of at least 3 months.
3. has histologically or cytologically documented advanced (unresectable and/or metastatic) solid tumor. Part 1A: recommend that participants have archival tissue not more than 3 years old. Part 1B and Part 2: participant has locally confirmed Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) tumor. Participant must have archival tumor tissue (not more than 3 years old) for retrospective confirmation of MSI-H or dMMR tumor by a central laboratory.
4. In Part 1A, has received and then progressed after or is intolerant to at least 1 standard treatment regimen in the advanced setting. The participant does not have alternative therapeutic options per PI's medical judgement. Preference should be given to: (1) participants with MSI-H or dMMR cancers that have progressed after checkpoint inhibitor (CPI) therapy and (2) participants with microsatellite stable cells (MSS) cancers that have progressed following at least one regimen of platinum, alkylating or topoisomerase containing chemotherapy.
5. has measurable disease at baseline according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by the PI.
6. has an Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.
7. has an adequate organ and marrow function.

Key Exclusion Criteria:

1. has not recovered (i.e., to Grade ≤ 1 or to baseline) from prior anti-cancer therapy-induced adverse events (AEs).
2. has received prior treatment with Werner (WRN) inhibitor.
3. has a history of relevant drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients, history of serious allergic reactions leading to hospitalization, or any other allergic reaction in general.
4. In Parts 1B and Part 2 Rescue: diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
5. has known additional malignancy that is progressing or has required active treatment within the past 3 years.
6. has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (ie, without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during the study screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of study treatment.
7. has mean resting QTcF > 470 ms (men and women) obtained from triplicate electrocardiograms (ECGs).
8. has active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Participants may enroll with the following conditions: Type 1 diabetes, hypothyroidism requiring hormone replacement, or skin disorders (vitiligo, psoriasis, or alopecia not requiring systemic treatment).
9. has history of (non-infectious) pneumonitis/pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
10. has active tuberculosis.
11. has any active infections requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) - Part 1 | 21 Days
  A DLT is a protocol-defined adverse event occurring during the DLT observation period.
Adverse Events (AEs) - Part 1 and Part 2 | From the time of first dose of study medication through 30 days following cessation of study treatment.
  Number of participants reporting adverse events or serious adverse events.

SECONDARY OUTCOMES:
Objective Response (OR) - Part 1 and Part 2 | Through study completion, an average of 2 years.
  OR defined as participants who have a complete response [CR] or partial response [PR] by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 as assessed by the Investigator.
Duration of Response (DOR) - Part 1 and Part 2 | Through study completion, an average of 2 years.
  DOR (defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first, in participants demonstrating CR or PR) by RECIST 1.1 as assessed by the Investigator.
Disease Control (DC) - Part 1 and Part 2 | Through study completion, an average of 2 years.
  DC defined as participants with a best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD) by RECIST 1.1 as assessed by the Investigator.
Progression-free survival (PFS) - Part 2 | Through study completion, an average of 2 years.
  PFS defined as the time from randomization to the first documented disease progression by RECIST 1.1 as assessed by the Investigator or death due to any cause, whichever occurs first.
Pharmacokinetic (PK) parameters of EIK1005 - AUC0-24 (Part 1 and Part 2) | Up to 1 year
  AUC0-24 (Area Under the plasma Concentration versus time curve from 0 to 24 hours): Measures total drug exposure over the first 24 hours after dosing of EIK1005 as monotherapy and in combination with pembrolizumab.
Pharmacokinetic (PK) parameters of EIK1005 - AUCtau,ss (Part 1 and Part 2) | Up to 1 year
  AUCtau,ss [Area Under the plasma Concentration versus time curve over one dosing interval (tau) at steady state]: Reflects average drug exposure during each dosing interval once the steady state has been reached for EIK1005 as monotherapy and in combination with pembrolizumab.
Pharmacokinetic (PK) parameters of EIK1005 - Cmax (Part 1 and Part 2) | Up to 1 year
  Cmax (Maximum Plasma Concentration) after dose administration of EIK1005 as monotherapy and in combination with pembrolizumab.
Pharmacokinetic (PK) parameters of EIK1005 - tmax (Part 1 and Part 2) | Up to 1 year
  tmax (the time required for the plasma concentration of the drug to reach maximum concentration after dose administration) of EIK1005 as monotherapy and in combination with pembrolizumab.
Pharmacokinetic (PK) parameters of EIK1005 - t½ (Half-life) (Part 1 and Part 2) | Up to 1 year
  Half-life (the time required for the plasma concentration of the drug to decrease by 50% after the dose administration) of EIK1005 as monotherapy and in combination with pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Nilou Mobashery, MD, Study Director — Eikon Therapeutics, Inc.
Locations (8):
- United States (3):
  - Morristown Medical Center, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Illawarra Cancer Care Centre (ICCC), Wollongong, New South Wales
  - Chris O'Brien Lifehouse (Sydney Cancer Centre), Camperdown, Victoria
  - Peninsula and Southeast Oncology (PASO) Medical, Frankston, Victoria
  - Olivia Newton John Cancer Research Institute, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Yes